CLINICAL TRIAL: NCT03785171
Title: Multimodal Magnetic Resonance Imaging Predicting Outcome After Surgical Revascularization in Patients With Moyamoya Disease
Brief Title: Predicative Value of Multimodal MRI in Moyamoya Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Xin Lou, Deputy Director of Department of Radiology, Chinese PLA General Hospital
Other Study IDs: Multimodal MRI-Moyamoya
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Moyamoya Disease; Magnetic Resonance Imaging
MeSH Terms: conditions — Moyamoya Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Moyamoya disease: The cohort includes patients with Moyamoya disease diagnosed by DSA examination who are treated by surgical revascularization.
  Interventions: Procedure: surgical revascularization

INTERVENTIONS:
Procedure: surgical revascularization — Indirect revascularization procedure

SUMMARY:
Moyamoya disease (MMD) is a nonatherosclerotic cerebrovascular abnormality, characterized by a progressive stenosis or occlusion of the intracranial internal carotid arteries (ICAs) and their proximal branches, with subsequent formation of collateral vessels ("puff of smoke"). In some cases, the posterior circulation can also be involved. MMD has been discovered around the world, but Asians carry the most possibility to develop this disease. Current treatment designed to prevent strokes by improving blood flow to the affected cerebral hemisphere including medical therapy and surgery. In particular, surgery included two general methods: direct and indirect revascularization. Compared with direct bypass, indirect procedures are more technically accessible and may reduce the possibility of complications, such as hyperperfusion. In addition, magnetic resonance imaging (MRI) with derived parameters have shown great potential in evaluating perfusion in patients, and could possibly predict surgical outcome. However, there is still lack of evidence of the predictive value of MRI in evaluating clinical and angiography improvement in patients with MMD.

DETAILED DESCRIPTION:
Imaging protocols:

3D TOF 3SLAB; SWAN; 3D ASL 2.0s; T1; T2; T2 Flair; DWI; tASL 2.0s; DCE; APT-CEST

Imaging evaluation:

1. Transfer contrast volume value measured by DCE;
2. ASL shows CBF in associated regions;
3. Stoke area measured by DWI and Flair;
4. PH values reflected by APT-CEST.

Treatment:

Surgery-indirect revascularization

Follow-up:

Baseline (MRI+DSA); 3-months follow-up (MRI); 6-months follow-up (MRI+DSA)

ELIGIBILITY:
Inclusion Criteria:

* DSA/MRA shows stenosis or occlusion in the distal internal carotid artery or the proximal portion of anterior/middle cerebral artery;
* Abnormal vascular network appeared in the brain;
* With the onset of cerebral ischemia/hemorrhage/TIA;
* No cerebral infarction or cerebral hemorrhage occurred within the last month;
* All MRI examination performed according to study protocol;
* Signed informed consent obtained from the patient or patient's legally authorized representative;
* Having complete medical history and clinical follow up;
* Imaging data can be processed.

Exclusion Criteria:

* Patients with moyamoya syndrome secondary to systemic diseases such as arteriosclerosis, sickle cell anemia, radiation therapy, etc.;
* Patients with severe mental disorders such as psychosis, liver and kidney dysfunction, poor blood pressure or blood glucose control, severe depression and substance abuse, low IQ, and acute phase of severe stroke with definite limb dysfunction should also be excluded.
* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Moyamoya disease
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-09-07 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Patients selection/stratification | Three months to 6 months
  Finding the effect of imaging biomarkers/patterns to provide therapy decision support

SECONDARY OUTCOMES:
Surgical outcome | Three months to 6 months
  Finding the effect of imaging biomarkers/patterns to reflect modified Rankin scale
Surgical response | Three months to 6 months
  Finding the effect of imaging biomarkers/patterns to reflect revascularized blood flow

CONTACTS AND LOCATIONS:
Overall Officials: Xin Lou, MD, Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided